CLINICAL TRIAL: NCT02926677
Title: Child Characteristics, Neuromarkers, and Intervention Components Impacting Treatment Outcome: A Randomized Controlled Trial of Cue-Centered Treatment (CCT), Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT), and Treatment as Usual (TAU)
Brief Title: Child Characteristics, Neuromarkers, and Intervention Components Impacting Treatment Outcome: CCT, TF-CBT, TAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Stanford Youth Solutions (Other); Drexel University (Other); Iowa State University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Victor G. Carrion, Professor-Med CTR LIne, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36092
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Child Trauma; Cue-Centered Treatment; Trauma-Focused Cognitive-Behavioral Therapy; fNIRs; CCT; TF-CBT; Posttraumatic stress; NIRX
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cue-Centered Therapy (CCT) (Experimental): Cue-Centered Therapy provides 15 sessions of treatment. Focuses on developing skills in recognizing stress cues and coping skills. Taught to self-soothe without the active involvement of a guardian. Teaches emotional, cognitive, and physiological conditioning to deal with ongoing traumatic stress. Will have a fNIR (NIRScout) scan at 4 time points throughout study (baseline, midpoint, end of treatment, and 3 month post-treatment)
  Interventions: Behavioral: Cue-Centered Treatment (CCT); Device: NIRScout
- Trauma-Focused CBT (TF-CBT) (Experimental): Trauma-Focused CBT provides 15 sessions of treatment. Focuses on reframing subconscious thought and emotions with emotional and cognitive conditioning. Uses the active involvement and support of guardians. Addresses discrete traumatic incidents in the past. Will have a fNIR (NIRScout) scan at 4 time points throughout study (baseline, midpoint, end of treatment, and 3 month post-treatment)
  Interventions: Behavioral: Trauma-Focused CBT (TF-CBT); Device: NIRScout
- Treatment as Usual (TAU) (Experimental): TAU is the current Standard treatment at Stanford Youth Solutions will serve as the control. The treatment is known as flexible integrated services. Will have a fNIR (NIRScout) scan at 4 time points throughout study (baseline, midpoint, end of treatment, and 3 month post-treatment)
  Interventions: Behavioral: Treatment as Usual; Device: NIRScout

INTERVENTIONS:
Behavioral: Cue-Centered Treatment (CCT) — Identify stress reactions and develop coping skills to deal with them independently. Helps address ongoing traumatic stressors.
  Arms: Cue-Centered Therapy (CCT)
Behavioral: Trauma-Focused CBT (TF-CBT) — Identifies negative cognitive/emotional patterns and helps re-frame them. Uses active support from guardians and focuses on emotional and cognitive conditioning. Focuses on discrete past incidents.
  Arms: Trauma-Focused CBT (TF-CBT)
Behavioral: Treatment as Usual — The control group. The standard treatment utilized at Stanford Youth Solutions
  Arms: Treatment as Usual (TAU)
Device: NIRScout — The device is a portable Functional Near-Infrared Spectroscopy (fNIRS) recording unit. NIRS technology uses specific wavelengths of light, introduced at the scalp to enable the non-invasive measurement of changes in the relative ratios of deoxygenated hemoglobin (deoxy-Hb) and oxygenated hemoglobin (oxy-Hb) in the capillary beds during brain activity.

SUMMARY:
This study is designed to examine three treatment conditions for traumatized youth: Cue-Centered Treatment (CCT), Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT), and Treatment as Usual (TAU) to determine which treatment works most effectively for which youth. The investigators would like to determine feasibility of training on the treatment interventions. In addition, this study aims to inform development of systems of care for chronically traumatized youth.

The investigators hope to determine whether 1) TF-CBT and CCT will have better outcomes than TAU, 2) Child characteristics predict better outcome in either TF-CBT or CCT and to identify which phases of treatment are most effective, and 3) Imaging findings will be predictors of improved outcome. This research is important because while there are many existing trauma interventions for youth, little is known about what is most essential in those interventions. This study will shed light on what components of treatment are most effective. Furthermore, there are minimal guidelines on how to select the most appropriate intervention for a particular child. This study will contribute to that knowledge by informing which interventions are suited best for which youth.

DETAILED DESCRIPTION:
The children will be referred from Stanford Youth Solutions and University of California, San Francisco. Caregivers will undergo a telephone screening according to the inclusion and exclusion criteria. Written consent for participation will be obtained from participants, parents and/or legal guardians. Participants will be randomly assigned to one of three treatment conditions: TF-CBT, CCT, or TAU. Assessments will be administered at 4 time points: 1) pre-treatment, 2) mid-therapy, 3) post-treatment, and 4) three month follow-up. A medical/developmental history form will be completed only pre-treatment. The UCLA PTSD Reaction Index (PTSD-RI) parent and child versions will be used to assess exposure to traumatic events and post-traumatic stress symptoms. Given that trauma has high comorbidity with depression and anxiety disorders these symptoms will be assessed using the Multidimensional Anxiety Scale for Children (MASC) and Children's Depression Inventory (CDI). Executive functioning will be assessed by both child and parent report using the Behavioral Rating Inventory of Executive Function (BRIEF).

In addition, functional near-infrared spectroscopy (fNIRs) will be conducted at each of these time points to assess tasks of working memory, response inhibition, and facial recognition. The investigators will be using the NIRScout which is a portable NIRS recording unit. NIRS technology uses specific wavelengths of light, introduced at the scalp, to enable the noninvasive measurement of changes in the relative ratios of deoxygenated hemoglobin (deoxy-Hb) and oxygenated hemoglobin (oxy-Hb) in the capillary beds during brain activity.

ELIGIBILITY:
Inclusion Criteria:

1. Exposure to at least one traumatic event and endorsement of any trauma symptoms on the UCLA PTSD Reaction Index for DSM-V
2. Ages 7-18
3. Willingness to participate in therapy and fNIRs imaging
4. Caregiver willing to participate in the study
5. Perpetrator of the traumatic event is not living in the home with the child

Exclusion Criteria:

1. Low cognitive functioning (IQ less than 70)
2. Substance dependence as defined by DSM criteria
3. Autism/Schizophrenia
4. Clinically significant medical illness

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor G Carrion, M.D., Principal Investigator — Stanford University; Hilit Kletter, PhD, Study Director — Stanford University; Flint Espil, PhD, Study Director — Stanford Univeristy
Locations (2):
- United States (2):
  - Stanford Youth Solutions, Sacramento, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cue-Centered Treatment (CCT): Cue-Centered Therapy provides 15 sessions of treatment. Focuses on developing skills in recognizing stress cues and coping skills. Taught to self-soothe without the active involvement of a guardian. Teaches emotional, cognitive, and physiological conditioning to deal with ongoing traumatic stress. Will have a fNIR (NIRScout) scan at 4 time points throughout study (baseline, midpoint, end of treatment, and 3 month post-treatment)
  Cue-Centered Treatment (CCT): Identify stress reactions and develop coping skills to deal with them independently. Helps address ongoing traumatic stressors.
  NIRScout: The device is a portable Functional Near-Infrared Spectroscopy (fNIRS) recording unit. NIRS technology uses specific wavelengths of light, introduced at the scalp to enable the non-invasive measurement of changes in the relative ratios of deoxygenated hemoglobin (deoxy-Hb) and oxygenated hemoglobin (oxy-Hb) in the capillary beds during brain activity.
Period: Overall Study
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Started | 25 | 22 | 26
Completed | 8 | 8 | 6
Not Completed | 17 | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 25 | 22 | 26 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.52 (3.00) | 13.41 (3.29) | 13.04 (3.05) | 12.97 (3.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 16 | 46
  Male | 8 | 9 | 10 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 1 | 4
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 5 | 8 | 6 | 19
  White | 15 | 11 | 15 | 41
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 26 | 73
UCLA Posttraumatic Stress Disorder (PTSD) Reaction Index for DSM 5 (child self-report) [Mean (Standard Deviation); unit: units on a scale] — The UCLA PTSD Reaction Index for DSM 5 is a 31 item self-report measure with child and parent versions. The total severity score ranging from 0-80 is obtained by summing the four symptom category sub-scales (criteria B, C, D, & E). The higher the score, the greater the PTSD severity. The items map onto the DSM 5 criteria for PTSD as well as assessing for dissociative subtype.
  units on a scale | 35.28 (15.66) | 37.10 (15.53) | 38.08 (14.04) | 36.80 (14.90)
UCLA Posttraumatic Stress Disorder (PTSD) Reaction Index for DSM 5 (parent report) [Mean (Standard Deviation); unit: units on a scale] — The UCLA PTSD Reaction Index for DSM 5 is a 31 item self-report measure with child and caregiver versions. The total severity score ranging from 0-80 is obtained by summing the four symptom category sub-scales (criteria B, C, D, & E). The higher the score, the greater the PTSD severity. The items map onto the DSM 5 criteria for PTSD as well as assessing for dissociative subtype.
  units on a scale | 31.13 (16.01) | 32.55 (13.73) | 33.92 (15.61) | 32.55 (15.02)
Multidimensional Anxiety Scale for Children (MASC 2) [Mean (Standard Deviation); unit: units on a scale] — The MASC 2 is a 50 item self-report measure assessing anxiety in the following sub-scales: separation anxiety/phobias, social anxiety, generalized anxiety, OCD, physical symptoms and harm avoidance. The total raw score is obtained by summing all the sub-scales. Total raw scores range from 0-150 with higher scores indicative of more severe anxiety. The raw score gets converted into a T-score interpreted as such: 45-55 average, 56-60 slightly above average, 61-65 above average, 66-70 much above average, and score of 70 or above is considered to be indicative of clinical anxiety.
  units on a scale | 63.76 (21.32) | 58.70 (24.25) | 59.56 (23.57) | 60.64 (22.84)
Children's Depression Inventory (CDI 2) [Mean (Standard Deviation); unit: units on a scale] — The CDI 2 is a 28 item self-report measure that assesses depressive symptoms in the past two weeks. Each item is scored from 0-2 and all items are summed to obtain the total score (total score range: 0-54; a score of 19 or higher is suggestive of clinical depression). The survey contains questions related to negative mood, negative self-esteem, interpersonal problems, anhedonia, and ineffectiveness.
  units on a scale | 17.38 (10.02) | 18.29 (9.93) | 17.42 (8.85) | 17.68 (9.42)
Behavior Rating Inventory of Executive Function (parent report) (BRIEF) [Mean (Standard Deviation); unit: units on a scale] — The BRIEF has 86 items that assess executive function with symptoms rated on a scale of 1-3. There are 8 clinical sub-scales (Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor) and two validity scales (Inconsistency and Negativity). A Global Executive Composite score (range 0-258 with higher scores indicative of greater impairment in executive function) is obtained by summing all 8 clinical sub-scales. The Global Executive Composite is converted to a T-score with T-scores of 65 or above considered in the clinical range.
  units on a scale
    Inhibit subscale | 18.35 (5.71) | 18.27 (5.95) | 17.75 (4.99) | 18.12 (5.47)
    Shift subscale | 15.87 (3.89) | 15.64 (3.33) | 15.87 (3.14) | 15.80 (3.42)
    Emotional Control subscale | 21.26 (4.18) | 21.45 (5.41) | 20.50 (4.87) | 21.06 (4.78)
    Initiate subscale | 15.65 (4.40) | 16.77 (2.65) | 16.79 (3.97) | 16.41 (3.75)
    Working Memory subscale | 20.39 (5.32) | 20.59 (5.00) | 20.79 (4.95) | 20.59 (5.02)
    Plan/Organize subscale | 22.65 (5.97) | 25.23 (5.41) | 23.96 (6.64) | 23.93 (6.05)
    Organization of Materials subscale | 12.83 (3.77) | 14.73 (2.75) | 13.42 (3.65) | 13.64 (3.47)
    Monitor subscale | 15.61 (3.96) | 16.32 (4.22) | 16.08 (3.69) | 16.00 (3.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in UCLA Posttraumatic Stress Disorder (PTSD) Reaction Index for DSM 5 (Child Self-report)
Description: The UCLA PTSD Reaction Index for DSM 5 is a 31 item self-report measure with child and caregiver versions. The total severity score ranging from 0-80 is obtained by summing the four symptom category sub-scales (criteria B, C, D, & E). A higher score corresponds to greater PTSD severity. The items map onto the DSM 5 criteria for PTSD as well as assessing for dissociative subtype.
Time Frame: Baseline and month 3 (end of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 6
score on a scale | -13.3 (12.1) | -17.8 (15.8) | -9.8 (10.2)

2. Primary Outcome: Change From Baseline in UCLA Posttraumatic Stress Disorder (PTSD) Reaction Index for DSM 5 (Parent Report)
Description: The UCLA PTSD Reaction Index for DSM 5 is a 31 item self-report measure with child and caregiver versions. Scores range from 0 to 80 (higher score indicates more sever PTSD symptoms). The items map onto the DSM-V criteria for PTSD as well as assessing for dissociative subtype.
Time Frame: Baseline and month 3 (end of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 6
score on a scale | -11.2 (11.1) | -17.4 (16.1) | -2.3 (10.2)

3. Secondary Outcome: Change From Baseline in Children's Depression Inventory (CDI 2)
Description: The CDI 2 is a 28 item self-report measure that assesses depressive symptoms in the past two weeks. Each item is scored from 0-2 and all items are summed to obtain the total score (total score range: 0-54; a score of 19 or higher is suggestive of clinical depression). The survey contains questions related to negative mood, negative self-esteem, interpersonal problems, anhedonia, and ineffectiveness.
Time Frame: Baseline and month 3 (end of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 6
score on a scale | -3.6 (7.3) | -4.7 (7.1) | -6.0 (9.6)

4. Secondary Outcome: Change From Baseline in Multidimensional Anxiety Scale for Children (MASC 2)
Description: The MASC 2 is a 50 item self-report measure assessing anxiety in the following sub-scales: separation anxiety/phobias, social anxiety, generalized anxiety, OCD, physical symptoms and harm avoidance. The total raw score is obtained by summing all the sub-scales. Total raw scores range from 0-150 with higher scores indicative of more severe anxiety. The raw score gets converted into a T-score interpreted as such: 45-55 average, 56-60 slightly above average, 61-65 above average, 66-70 much above average, and score of 70 or above is considered to be indicative of clinical anxiety.
Time Frame: Baseline and month 3 (end of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 6
score on a scale | -15.8 (20.5) | -12.8 (11.2) | -16.8 (28.7)

5. Secondary Outcome: Change From Baseline in the Behavior Rating Inventory of Executive Function (BRIEF) (Parent Report)
Description: The BRIEF is an 86 item measure that assesses impairment in executive function with symptoms rated on a likert scale of 1 "never", 2 "sometimes" or 3 "often". There are 8 clinical sub-scales (Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor) and two validity scales (Inconsistency and Negativity). A Global Executive Composite score is obtained by summing all 8 clinical sub-scales. The Global Executive Composite ranges from 0-258 with higher scores indicating greater impairment in executive functions. The Global Executive Composite gets converted to a T-score with T-scores of 65 or above considered in the clinical range.
Time Frame: Baseline to month 3 (end of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cue-Centered Therapy (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 6
score on a scale
  Inhibit subscale | 2.22 (1.72) | 0.44 (4.25) | -2.00 (5.73)
  Shift subscale | 0.56 (1.67) | 2.33 (2.24) | -0.83 (4.36)
  Emotional Control subscale | 2.56 (3.28) | 3.89 (2.85) | 0.17 (4.12)
  Initiate subscale | 1.11 (3.14) | 1.11 (2.71) | 1.17 (2.64)
  Working memory subscale | 2.67 (2.29) | 2.00 (3.35) | -0.33 (4.23)
  Plan/Organize subscale | 1.78 (3.03) | 2.22 (5.45) | -0.67 (4.59)
  Organization of Materials subscale | 1.00 (3.12) | 1.44 (1.74) | 1.00 (2.00)
  Monitor subscale | 0.78 (2.44) | 0.44 (3.32) | -2.17 (5.46)

ADVERSE EVENTS:
Time Frame: Up to 4 1/2 months
Arm/Group | Cue-Centered Treatment (CCT) | Trauma-Focused CBT (TF-CBT) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/26

LIMITATIONS AND CAVEATS:
The study was underpowered because the number of participants with analyzable data did not meet the threshold for the planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT02926677/ICF_000.pdf
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT02926677/Prot_001.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT02926677/SAP_002.pdf